CLINICAL TRIAL: NCT04468425
Title: Open-label, Fixed-sequence, Two-period Comparative Bioavailability Study of Tofacitinib From Repeated Topical Applications of Tofacitinib Citrate Topical Gel 3.2% to Single Oral Administration of Xeljanz 5 mg Tablet in Healthy Subjects
Brief Title: Tofacitinib Citrate Topical Gel 3.2% FDA BA Bridging Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TWi Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: AC-1101-PK-001
Record Dates: First submitted 2020-07-07; First posted 2020-07-13 (Actual); Last update posted 2021-11-29 (Actual); Status verified 2021-11

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — tofacitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pharmacokinetic Study (Experimental): Period 1 (Day 1) and 2 (Day 8 - Day 21) separated by 7-day washout period. Period 1: A single 5 mg tofacitinib tablet will be administered orally on Day 1.
  Period 2: Repeat dosing of Tofacitinib Citrate Topical Gel 3.2% to approximately 10% BSA in the morning of Day 8 and twice daily from Day 9 to Day 20 with the last dose in the morning of Day 21.
  Interventions: Drug: Tofacitinib Citrate

INTERVENTIONS:
Drug: Tofacitinib Citrate — Period 1: Xelijanz® 5 mg tablet (tofacitinib citrate) for single oral dosing. Period 2: Tofacitinib Citrate Topical Gel 3.2% for repeat topical dosing BID for 14 days.

SUMMARY:
This is a Phase 1, single center, open-label, fixed sequence, two-period pharmacokinetic (PK) study to evaluate the safety and relative systemic bioavailability of topical and oral tofacitinib formulations in approximately 14 healthy subjects. Participants will receive a single oral dose of tofacitinib 5 mg tablet in Period 1 of the study followed by a 7-day washout period. In Period 2, participants will receive repeat administration of Tofacitinib Citrate Topical Gel 3.2% BID for 14 days.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, smoker (no more than 25 cigarettes or equivalent daily) or non-smoker, ≥18 and ≤60 years of age, with BMI >18.5 and <30.0 kg/m2 and body weight ≥50.0 kg for males and ≥45.0 kg for females.
2. Healthy as defined by:

   1. The absence of clinically significant illness. Subjects vomiting within 24 hours pre dose will be carefully evaluated for upcoming illness/disease. Inclusion pre dosing is at the discretion of the Investigator;
   2. The absence of clinically significant history of dermatological, neurological, endocrine, cardiovascular, respiratory, hematological, immunological, psychiatric, gastrointestinal, renal, hepatic, and metabolic disease.
3. Females of childbearing potential who are sexually active with a male partner must be willing to use one of the following acceptable contraceptive methods throughout the study and for 30 days after the last study drug administration:

   1. Intra-uterine contraceptive device without hormone release system placed at least 4 weeks prior to study drug administration;
   2. Male condom with intravaginally applied spermicide started at least 21 days prior to study drug administration;
   3. Sterile male partner (vasectomized since at least 6 months).
4. Absence of excessive body hair at the topical application site, or willing to have excess body hair removed prior to dosing.
5. Capable of consent.

Exclusion Criteria:

1. Presence of any clinically significant abnormality at physical examination, clinically significant abnormal laboratory assessment or positive test for hepatitis B, hepatitis C, or HIV found during medical screening.
2. Positive urine drug screen or alcohol breath test at screening.
3. History of allergic reactions to tofacitinib or other related drugs, or to any excipient in the formulation.
4. Positive pregnancy test at screening.
5. Clinically significant ECG abnormalities or vital sign abnormalities (systolic blood pressure lower than 90 or over 140 mmHg, diastolic blood pressure lower than 50 or over 90 mmHg, or heart rate less than 50 or over 100 bpm) at screening.
6. History of significant alcohol abuse within 1 year prior to screening or regular use of alcohol within 6 months prior to the screening visit (more than 14 units of alcohol per week [1 unit = 150 mL of wine, 360 mL of beer, or 45 mL of 40% alcohol]).
7. History of significant drug abuse within 1 year prior to screening or use of soft drugs (such as marijuana) within 3 months prior to the screening visit or hard drugs (such as cocaine, phencyclidine [PCP], crack, opioid derivatives including heroin, and amphetamine derivatives) within 1 year prior to screening.
8. Participation in a clinical research study involving the administration of an investigational or marketed drug or device within 30 days prior to the first dosing, administration of a biological product in the context of a clinical research study within 90 days prior to the first dosing, or concomitant participation in an investigational study involving no drug or device administration.
9. Use of medications for the timeframes specified below, with the exception of medications exempted by the Investigator on a case-by-case basis because they are judged unlikely to affect the pharmacokinetic profile of the study drug or subject safety e.g. topical drug products without significant systemic absorption (not including topical drug products administered to the gel application site):

   1. Prescription medications within 14 days prior to the first dosing;
   2. Over-the-counter products and natural health products (including herbal remedies, homeopathic and traditional medicines, probiotics, food supplements such as vitamins, minerals, amino acids, essential fatty acids, and protein supplements used in sports) within 7 days prior to the first dosing, with the exception of the occasional use of acetaminophen (up to 2 g daily);
   3. Depot injection or implant of any drug within 3 months prior to the first dosing;
   4. Any drugs known to induce or inhibit hepatic drug metabolism via the CYP3A4 and CYP2C19 enzymes within 30 days prior to first dose;

      * Examples of inducers for CYP3A4 include barbiturates, carbamazepine, phenytoin, glucocorticoids, St. John's wort, etc.
      * Examples of inhibitors for CYP3A4 include HIV antivirals, clarithromycin, ciprofloxacin, gestodene, etc.
      * Examples of inducers for CYP2C19 include carbamazepine, norethindrone, prednisone, rifampicin, etc.
      * Examples of inhibitors for CYP2C19 include proton pump inhibitors, fluoxetine, ketoconazole, etc.
10. Donation of plasma within 7 days prior to dosing. Donation or loss of blood (excluding volume drawn at screening) of 50 mL to 499 mL of blood within 30 days, or more than 499 mL within 56 days prior to the first dosing.
11. Breast-feeding subject.
12. History of active tuberculosis or exposure to endemic areas within 8 weeks prior to QuantiFERON®-TB testing performed at screening.
13. Positive QuantiFERON®-TB indicating possible tuberculosis infection.
14. Immunization with a live attenuated vaccine within 1 month prior to dosing or planned vaccination during the course of the study.
15. History of clinically significant opportunistic infection e.g. invasive candidiasis or pneumocystis pneumonia.
16. Serious local infection e.g. cellulitis, abscess, or systemic infection e.g. septicemia, within 3 months prior to screening.
17. Presence of fever (body temperature >37.6 °C) e.g. a fever associated with a symptomatic viral or bacterial infection, within 2 weeks prior to the first dosing.
18. Presence of sunburn at the gel application site, or excessive exposure to ultraviolet light such as sunlight or a tanning lamp, or recent use of laser at the gel application areas that would prevent a safe application of the gel formulation as judged by the Investigator, within 7 days before the gel application.
19. Presence of tattoos or significant skin aberrations at the gel application site, which in the opinion of the investigator, would interfere with the ability to perform an accurate dermal reaction assessment.
20. Any reason that, in the opinion of the Investigator, would prevent the subject from participating in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2020-12-21 (Actual); Study Completion 2020-12-21 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration [Cmax] of tofacitinib from single oral dosing in Period 1 | Day 1
Area Under Curve [AUC] of tofacitinib from single oral dosing in Period 1 | Day 1
Maximum Plasma Concentration [Cmax] of tofacitinib from repeat topical dosing in Period 2 | Day 8
Area Under Curve [AUC] of tofacitinib from repeat topical dosing in Period 2 | Day 8
Maximum Plasma Concentration [Cmax] of tofacitinib from repeat topical dosing in Period 2 | Day 21
Area Under Curve [AUC] of tofacitinib from repeat topical dosing in Period 2 | Day 21
Safety and tolerability of Tofacitinib Citrate Topical Gel 3.2% as assessed by treatment-emergent adverse events and Dermal Reaction Scoring, respectively. | Day 24

CONTACTS AND LOCATIONS:
Locations (1):
- Syneos Health Facility, Québec, Canada

IPD SHARING:
Plan to Share IPD: No